CLINICAL TRIAL: NCT06554873
Title: Adaptive Use of Nicotine Substitution to Maintain Smoking Reduction/Abstinence in Nicotine Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Global Action to End Smoking (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATS2
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation; Harm Reduction
MeSH Terms: conditions — Smoking Cessation; Harm Reduction | interventions — Nicotine; Tobacco Use Cessation Devices; Nicotine Chewing Gum; Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nicotine Non-Responders (Experimental): Participants that were not successful in reducing their expired carbon monoxide by the end of week 2 will not continue in the study.
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product; Other: NJOY e-cigarette; Other: on!
- Nicotine Responders - Group 1 (Experimental): Participants that were successful in reducing their expired carbon monoxide by the end of week 2 will be randomized to continued use of their choice of nicotine products for an additional 10 weeks (12-week total treatment period).
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product; Other: NJOY e-cigarette; Other: on!
- Nicotine Responders - Group 2 (Experimental): Participants that were successful in reducing their expired carbon monoxide by the end of week 2 will be randomized to continued use of their choice of nicotine products for an additional 22 weeks (24-week total treatment period).
  Interventions: Drug: Nicoderm; Drug: Nicorette 4Mg Chewing Gum; Drug: Nicorette Lozenge Product; Other: NJOY e-cigarette; Other: on!

INTERVENTIONS:
Drug: Nicoderm — Depending on responder status and group assignment the maximum amount of time nicotine patches will be used is 24 weeks. The final four weeks of nicotine patch treatment will comprise 2 weeks of 14 mg patches and two weeks of 7 mg patches.
  Other Names: Nicotine Patch
Drug: Nicorette 4Mg Chewing Gum — 4mg Nicorette gum (flavors - cinnamon surge, fruit chill, and mint); as needed maximum usage 24 weeks.
  Other Names: Nicotine gum
Drug: Nicorette Lozenge Product — 4mg Nicorette mint lozenge; as needed maximum usage 24 weeks.
  Other Names: Nicotine lozenge
Other: NJOY e-cigarette — Each NJOY Classic Tobacco and Menthol pod is pre-filled with 1.9 mL of e-liquid with 5% nicotine (by weight); as needed maximum usage 24 weeks.
Other: on! — 4mg on! Nicotine Pouch (flavors - Berry, Mint, and Original); as needed for maximum usage 24 weeks.
  Other Names: Nicotine pouch

SUMMARY:
To determine whether smokers who initially respond (within 2 weeks) to nicotine products (including nicotine replacement therapy, e-cigarettes, nicotine pouches) by reducing their smoking by ≥50% can be successfully maintained on use of these noncombustible nicotine alternatives to cigarettes for 6 months, and whether this results in sustained smoking reduction/abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult smoker of combustible cigarettes.
* Age 22 to 65 years at time of screening (verified by government issued ID).
* Smoke cigarettes for ≥12 months prior to screening.
* Currently smokes at least 10 tobacco cigarettes per day.
* Screening eCO ≥ 10 ppm.
* Voluntarily provides consent for participation by signing the informed consent form (ICF).
* Willing and able to comply with study requirements.

Exclusion Criteria:

* Unable to read, speak or understand English
* Has a history or presence of clinically significant medical or psychiatric disease, or any other condition that would in the PI's judgement jeopardize the safety of the participant, impair the participant's ability to comply with study procedures, or impact the validity of the study results.
* Has used nicotine-containing e-cigarettes (or vapes) or any nicotine replacement therapy (nicotine patch, nicotine gum, nicotine spray, nicotine inhaler, nicotine lozenge) or prescription smoking cessation medications, including, but not limited to, varenicline (Chantix*) or bupropion (Zyban®) within the past 30 days.

If female, participant is pregnant, nursing, or intends to become pregnant during the time period from screening through the end of study.

* Has participated in a research study about tobacco products or ENDS within the past 30 days.
* Has participated in a smoking cessation or nicotine switching research study in the past year.
* Smokes or vapes cannabis more than once a week.
* Cannabis Use Disorder Identification Test-Revised (CUDIT-R) score of 8 or greater.
* Heterosexually active participants of Childbearing Potential (not sterilized by tubal ligation, oophorectomy, hysterectomy, or other surgical methods, or post-menopausal) that do not agree to practice medically appropriate methods of birth control (or remain abstinent) during the course of the trial. Medically acceptable methods of birth control include: vasectomy, vaginal diaphragm with spermicide, intrauterine device, hormonal birth control (oral, injected, or implanted), condom with spermicide, or sponge with spermicide.
* Subgroup enrollment is complete.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence - CO | Week 12 and Week 24
  To determine whether maintained use of nicotine products can help sustain smoking abstinence rates for early responders. An expired air CO reading of ≤ 5 ppm at 24 weeks.

SECONDARY OUTCOMES:
Smoking abstinence - Self report of no smoking | Week 12 and Week 24
  Percent smoking abstinence at 12 weeks and 24 weeks, defined on an intent-to-treat basis as a self-report of no-smoking for the prior 7 days
Reduction in Expired Air CO | Week 12 and Week 24
  Percent of participants achieving a 50% reduction in expired air CO at 12 weeks and 24 weeks relative to baseline.
Usage of Nicotine Products | Week 1 through Week 24, Week 36
  Self-reported usage of nicotine products.
Saliva Cotinine Concentrations | Week 12, Week 24, Week 36
  Saliva cotinine concentrations reflective of nicotine product usage in smoking-abstinent individuals.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina